CLINICAL TRIAL: NCT02103452
Title: Edessy STEM CELL SCORE (ESS), Endometrium, Endometrioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, Professor, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17819555
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-03

CONDITIONS: Endometriosis, Ovarian
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ovarian endometrioma (Experimental): Ovarian and endometrial samples
  Interventions: Procedure: Ovarian and endometrial samples
- normal ovary (Experimental): Ovarian and endometrial samples
  Interventions: Procedure: Ovarian and endometrial samples

INTERVENTIONS:
Procedure: Ovarian and endometrial samples — Ovarian and endometrial samples were evaluated by hematoxlin &eosin for histopathology (HP) and of oct-4 for immunohistochemistry (IH) for SCE

SUMMARY:
Purpose of this study is to evaluate stem cell expression (SCE) in endometriotic (E) and non endometriotic ovarian and endometrial tissues.

DETAILED DESCRIPTION:
This study was conducted on 40 women at Al-Azhar University Hospitals. They are divided into two equal groups, group 1 with ovarian endometrioma and group 2 with normal ovary. Ovarian and endometrial samples were evaluated by hematoxlin & eosin for histopathology (HP) and of oct-4 for immunohistochemistry (IH) for SCE.

Evaluation of IH parameters revealed that the most important factors for evaluating SC were arranged as score ( Edessy Stem Cell Score=ESS).

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years and did not receive hormonal treatment for three month

Exclusion Criteria:

* Diabetes mellitus, cardiovascular and kidney diseases, adenomyosis, Uterine fibroid Endometrial carcinoma and Poly cystic ovary

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Edessy Stem Cell Score (ESS) | 1 week
  ESS
  * Intensity of stem cell marker: Negative to mild =0, Moderate =1, Strong =2
  * Percentage of stained cells: 0 =0, 0-50%= 1, >50-100% =2.
  * Focality : None =0, Focal =1, Diffuse= 2
  * Distribution: None= 0, Epithelial or mesenchymal= 1, Epithelial and mesenchymal= 2.
  * Localization of positive stained cell: None=0, Cytoplasmic or nuclear =1, Cytoplasmic and nuclear= 2

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, MD, Principal Investigator — Al-Azhar University; Hala hosni, MD, Study Director — Cairo University; Magdy Olama, MD, Study Director — Al-Azhar University; Mohammad A Sattar, MD, Study Chair — Al-Azhar University; Ahmad Monir, MSc, Study Chair — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Cairo Governorate, Egypt